CLINICAL TRIAL: NCT07350031
Title: Cortisol Assessment in Patients With Adrenal Incidentalomas
Brief Title: Serum and Salivary Cortisol Assessment in Patients With Adrenal Incidentalomas and Healthy Controls
Acronym: SALICOR
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Nanna Thurmann Jørgensen, MD, Rigshospitalet, Denmark
Other Study IDs: H-16041718
Record Dates: First submitted 2025-09-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Adrenal Incidentaloma; Hypercortisolism
Keywords: Salivary cortisol, DST, MACS, hypercortisolism, reference interval
MeSH Terms: conditions — Adrenal incidentaloma; Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with adrenal incidentalomas
  Interventions: Diagnostic Test: 1 mg overnight dexamethasone suppression test
- Healthy control group
  Interventions: Diagnostic Test: 1 mg overnight dexamethasone suppression test

INTERVENTIONS:
Diagnostic Test: 1 mg overnight dexamethasone suppression test — Included participants will undergo routine medical examination including 1 mg dexamethasone-suppression-test, 24 h urine sample, and measurement of plasma-adrenocorticotropin (ACTH). In addition to the routine biochemical tests, saliva samples will be collected the morning and evening before intake of dexamethasone as well as the following morning together with serum cortisol.

SUMMARY:
The goal of this observational study is to evaluate the diagnostic accuracy of salivary cortisol compared with serum cortisol after a 1 mg overnight dexamethasone suppression test in participants (N = 100) with adrenal incidentalomas and healthy control participants (N = 100). The main question it aims to answer is:

Are salivary cortisol and serum cortisol equal diagnostic tools for endogenous hypercortisolism?

The inclusion of healthy controls will serve as a reference population to define the central 95 % reference interval for the serum and salivary cortisol levels.

Participants will undergo routine medical examination of adrenal incidentalomas including 1 mg dexamethasone-suppression-test, 24 h urine sample, and measurement of plasma-adrenocorticotropin (ACTH). In addition to the routine biochemical tests, saliva samples will be collected the morning and evening before intake of dexamethasone as well as the following morning together with serum cortisol.

ELIGIBILITY:
Inclusion Criteria (patients):

* age ≥ 18 years, a new diagnosis of an adrenal incidentaloma (defined as an adrenal mass > 1 cm detected when using diagnostic imaging for non-related reasons).

Inclusion Criteria (controls):

* age ≥ 18 years, no previous history of conditions involving the adrenal glands

Exclusion Criteria (patients):

* active cancer; an adrenal incidentaloma suspected of malignancy; bilateral adrenal incidentalomas; pregnancy and breastfeeding; conditions or medical treatments that interfere with dexamethasone metabolism and cortisol metabolism/measurements; severe comorbidities; chronic kidney disease (defined as an estimated glomerular filtration rate < 60 ml/min); and inability to provide written informed consent.

Exclusion Criteria (controls):

* active cancer; pregnancy and breastfeeding; conditions or medical treatments that interfere with dexamethasone metabolism and cortisol metabolism/measurements; severe comorbidities; chronic kidney disease (defined as an estimated glomerular filtration rate < 60 ml/min); and inability to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient group were patients newly diagnosed with an adrenal incidentaloma and referred to either the Department of Nephrology and Endocrinology, Copenhagen University Hospital, Rigshospi-talet, Denmark or Department of Medicine, Copenhagen University Hospital Herlev Gentofte, Herlev, Denmark.
  The controls were recruited through social media, online participant recruitment platform , the hospital website, and physical posters in public spaces around Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol and cortisone in patients and controls following an overnight dexamethasone suppression test | Baseline (Day 0, 08:00-09:00 hour) and post-dexamethasone (Day 1, 08:00-09:00 hour)
  Cross-sectional evaluation of serum and salivary cortisol and cortisone after an overnight 1 mg dexamethasone suppression test in patients with adrenal incidentalomas and healthy controls.

IPD SHARING:
Plan to Share IPD: Undecided